CLINICAL TRIAL: NCT02517112
Title: 3D Ballistocardiography in Microgravity
Acronym: B3D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-126
Record Dates: First submitted 2015-07-23; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiovascular parameters measurements (Other)
  Interventions: Other: Parabolic flight; Other: Cardiovascular parameters measurements; Device: 3D-BCG sensor

INTERVENTIONS:
Other: Parabolic flight
Other: Cardiovascular parameters measurements — with Ballistocardiography (BCG), electric cardiography (ECG), impedance cardiography (ICG) and echocardiography
Device: 3D-BCG sensor

SUMMARY:
3-D Ballistocardiography (BCG) recording was performed in microgravity during the Spacelab D2 missions on a single astronaut. The results from this experiment have been published in the literature: the influence of respiration have been demonstrated and the signal processing methodology for the reconstruction of the displacement in one cardiac cycle have been developed. A 3D-BCG sensor has been developed and a collaboration to perform a sustained microgravity experiment onboard the Russian segment of ISS has been initiated. To be integrated in the PNEUMOCARD device, this new sensor needs to be tested in microgravity before implemented on ISS.

The aim of the present parabolic flight study is to serve as a feasibility demonstrator and test bed in order to evaluate the feasibility of 3D-BCG in sustained microgravity and to test whether the sensitivity of the developed 3D-BCG sensor is appropriate

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Whose 4 chamber view of the heart during a breath hold is easy to get during a routine cardiac echocardiography (M-Mode - apical view).
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Difficulty to obtain a clear echocardiography.
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Heart rate | baseline
  evaluated by BCG, ECG, ICG and echocardiography during the free-floating protocol
stroke volume | baseline
  evaluated by BCG, ECG, ICG and echocardiography during the free-floating protocol
ejection fraction | baseline
  evaluated by BCG, ECG, ICG and echocardiography during the free-floating protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France